CLINICAL TRIAL: NCT07285577
Title: Fractional Microneedling Radiofrequency Versus Facial Muscle Exercises for Facial Rejuvenation: A Randomized Controlled Trial
Brief Title: Facial Muscle Exercises vs Fractional Microneedling Radiofrequency for Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, heba ahmed abdelgayed ibrahim, Lecturer of Dermatology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-63-2022
Record Dates: First submitted 2025-12-10; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Facial Aging
Keywords: Facial rejuvenation; Fractional microneedling radiofrequency; Face yoga; Facial muscle exercises; Non-surgical facelift; Radiofrequency; Wrinkle reduction; Skin texture improvement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Facial Muscle Exercises (FME) (Experimental): Participants received an 8-week facial muscle exercise program consisting of weekly online sessions led by the investigator and daily home exercises. Exercises targeted nasolabial folds and jawline using techniques such as "Big O," "Nasolabial Lift Up," "Nasolabial Smoother," "Rolly Polly," "Swan Neck," and "Pulled Tongue," following the Face Yoga method.
  Interventions: Behavioral: Facial Muscle Exercise Program
- Fractional Microneedling Radiofrequency (FMR) (Experimental): Participants underwent three sessions of fractional microneedling radiofrequency using the Vivace® device at 4-week intervals. Non-insulated microneedles were used with parameters: depth 3.5 mm, power 8 W, pulse duration 800 ms. Local anesthetic cream applied before each session; topical antibiotics and moisturizers used post-procedure.
  Interventions: Device: Vivace® Fractional Microneedling Radiofrequency

INTERVENTIONS:
Behavioral: Facial Muscle Exercise Program — Eight-week course with weekly online sessions and daily home exercises demonstrated via video. Exercises aimed to improve facial muscle tone and lifting effect.
  Arms: Facial Muscle Exercises (FME)
Device: Vivace® Fractional Microneedling Radiofrequency — Three sessions spaced 4 weeks apart; non-insulated microneedles; depth 3.5 mm; power 8 W; pulse 800 ms; pre-treatment topical anesthesia; post-treatment care with antibiotics and moisturizers.
  Arms: Fractional Microneedling Radiofrequency (FMR)

SUMMARY:
This randomized controlled trial compared the effectiveness and safety of fractional microneedling radiofrequency (FMR) and facial muscle exercises (FME) for facial rejuvenation in females with mild to moderate facial aging. Forty participants aged 32-65 were randomized to either an 8-week FME program or three FMR sessions at 4-week intervals. Outcomes included modified quantitative comprehensive grading scale of aging (MQCGS), wrinkle severity rating scale (WSRS), physician global aesthetic improvement score (PGAI), subject global aesthetic improvement score (SGAIS), and patient satisfaction. Primary endpoints were treatment success (≥25% improvement in PGAI) and patient satisfaction at Day 90. Secondary outcomes assessed changes in aging scores, wrinkle severity, and improvement type (lifting versus texture effects). Ethics approval was obtained from the Research Ethics Committee, Faculty of Medicine, Cairo University.

DETAILED DESCRIPTION:
Facial aging involves changes in skin texture, loss of volume, and tissue descent. Fractional microneedling radiofrequency (FMR) delivers controlled thermal injury via microneedles to stimulate collagen and elastin, with proposed benefits for skin texture and firmness. Facial muscle exercises (FME), or face yoga, aim to strengthen facial muscles, enhance tone, and lift sagging tissues. This single-center, outpatient, randomized, active-controlled, parallel-group trial enrolled 40 female participants aged ≥30 years with mild to moderate facial aging. Group A received an 8-week FME program (weekly online sessions plus daily home exercises). Group B underwent three FMR sessions using Vivace® device (non-insulated microneedles, 3.5 mm depth, 8 W, 600 ms pulse) at 4-week intervals. Primary outcomes were treatment success (≥25% improvement in PGAI) and patient satisfaction at Day 90. Secondary outcomes included MQCGS, WSRS, SGAIS, and improvement type (lifting versus texture). The study aimed to compare the two interventions across these outcome measures. Ethics approval was granted by the Research Ethics Committee, Faculty of Medicine, Cairo University; informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged ≥30 years
* Mild to moderate facial aging (defined as grade 2-3 on Modified Quantitative Comprehensive Grading Scale of Aging and grade 2-4 on Wrinkle Severity Rating Scale)
* Literate and able to follow instructions
* Familiar with using online applications (e.g., Zoom) and have reliable internet access
* Provided written informed consent for participation and photography

Exclusion Criteria:

* Age <30 years
* Severe facial aging (grade 4 on MQCGS and grade 5 on WSRS)
* Current smoker
* History of previous facelift surgery or thread lifting Botulinum toxin or filler injection within the past 12 months
* Mesotherapy or topical rejuvenating therapy within the past 3 months
* Body dysmorphic disorder
* Medical history of autoimmune diseases, diabetes, or systemic conditions affecting healing
* Pregnancy or lactation
* Illiteracy or inability to follow instructions
* Lack of internet access or inability to use online applications

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study included female participants aged 30 years or older with mild to moderate facial aging.
Enrollment: 40 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Treatment Success (≥25% improvement in Physician Global Aesthetic Improvement Score) | Day 90 (End of Study)
  Proportion of participants achieving ≥25% improvement in PGAI compared to baseline.
Patient Satisfaction | Day 90 (End of Study)
  Measured on a 3-point scale (0 = not satisfied, 1 = moderately satisfied, 2 = very satisfied).

SECONDARY OUTCOMES:
Modified Quantitative Comprehensive Grading Scale of Aging (MQCGS) | Baseline, Day 30, Day 60, Day 90
  Change from baseline in Modified Quantitative Comprehensive Grading Scale of Aging (MQCGS) score. Scale range: 0-33 points, with higher scores indicating more severe facial aging (worse outcome).
Wrinkle Severity Rating Scale (WSRS) | Baseline, Day 30, Day 60, Day 90
  Change from baseline in Wrinkle Severity Rating Scale (WSRS) score for nasolabial folds. Scale range: 1-5, with higher scores indicating more severe wrinkles (worse outcome).
Subject Global Aesthetic Improvement Score (SGAIS) | Day 30, Day 60, Day 90
  Patient-reported improvement compared to baseline using Subject Global Aesthetic Improvement Score (SGAIS). Scale range: -1 to +3, with higher scores indicating greater improvement (better outcome). (-1 = worse, 0 = no change, +1 = improved, +2 = much improved, +3 = very much improved)
Improvement Type | Day 90
  Classification of improvement as "lifting," "texture," or "both" based on blinded dermatologist review.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Aini Hospital, Cairo, English (English), Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single-center study with a small sample size, and de-identification cannot be fully guaranteed. Aggregate results, including summary statistics and outcome analyses, will be made available through publication